CLINICAL TRIAL: NCT06922383
Title: A Phase 1b/2 Study of Arfolitixorin Combined With 5-fluorouracil, Oxaliplatin, and Bevacizumab in First-line Treatment of Metastatic Colorectal Cancer
Brief Title: A Clinical Study of Arfolitixorin in Patients With mCRC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISO-CC-010; 2024-516802-43-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: arfolitixorin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients in this study will receive the IMP arfolitixorin combined with 5-FU, oxaliplatin, and bevacizumab (ARFOX + bevacizumab). The other medications 5-FU, oxaliplatin, and bevacizumab, are also referred to as auxiliary medicinal products (AxMPs).
  In Phase 1b of the study, a dose escalation design will be utilized to identify the optimal dose and duration of administration of arfolitixorin to be used in combination with 5-FU, oxaliplatin and bevacizumab.
  The Phase 2 part of the study will be a randomized study where patients will be allocated to 1 of 2 dose levels of arfolitixorin. The higher dose level will be the maximum tolerated dose as determined in Phase 1b, and the lower dose level will be a dose level below the maximum tolerated dose as determined in Phase 1b, i.e., 1 of the dose levels as determined by the Safety Review Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose level (Experimental): The higher dose level of arfolitixorin in Phase 2 will be the maximum tolerated dose as determined in Phase 1b. The arfolitixorin will be given as i.v. infusion. Patients in this study will receive the IMP arfolitixorin combined with 5-FU, oxaliplatin, and bevacizumab (ARFOX + bevacizumab). The duration of the infusion will be determined in Phase 1b.
  Interventions: Drug: arfolitixorin (ARFOX + bevacizumab)
- Low dose level (Experimental): The lower dose level of arfolitixorin in Phase 2 will be a dose level below the maximum tolerated dose as determined in Phase 1b. The arfolitixorin will be given as i.v. infusion. Patients in this study will receive the IMP arfolitixorin combined with 5-FU, oxaliplatin, and bevacizumab (ARFOX + bevacizumab). The duration of the infusion will be determined in Phase 1b.
  Interventions: Drug: arfolitixorin (ARFOX + bevacizumab)

INTERVENTIONS:
Drug: arfolitixorin (ARFOX + bevacizumab) — Every 14 days during treatment phase, Bevacizumab will be administered as an i.v. infusion of 5 mg/kg, Oxaliplatin will be administered as an 85 mg/m2 i.v. infusion, 5-FU will be administered as a 400 mg/m2 i.v. bolus + a 2,400 mg/m2 i.v. infusion and Arfolitixorin will be administred as an i.v. infusion.

SUMMARY:
This is a clinical research study taking place in Germany. Patients with colorectal cancer at a stage of the disease where metastases occur may take part in the study. A maximum of 60 people will participate in the study.

There is already a standard therapy for treatment of colorectal cancer. This therapy contains a combination of the medicines leucovorin, fluorouracil, oxaliplatin and bevacizumab.

The sponsoring company is developing the new therapy called arfolitixorin. In this study, patients with colorectal cancer will be given arfolitixorin instead of the standard treatment leucovorin. Different patients will receive treatment with different strengths (doses) of arfolitixorin. Treatment with fluorouracil, oxaliplatin and bevacizumab will also be administrated.

The researchers want to find out if arfolitixorin could have an advantage over the standard therapy with leucovorin. They also want to investigate which dose of arfolitixorin is the most optimal dose to give to other patients and also to study if arfolitixorin is safe to use.

The product being tested, arfolitixorin, like leucovorin, belongs to a group of substances called folates which are naturally occurring forms of a type of B vitamin. Folates are administered in combination with one or more chemotherapeutic agents to enhance their effect on cancer cells.

The main mechanism of action of arfolitixorin is the same as that of leucovorin when used together with fluorouracil. However, leucovorin must first be converted into the active form in the body, whereas arfolitixorin already is in the active form. Leucovorin does not work equally well in all patients. By bypassing the metabolic activation of arfolitixorin, it is assumed that arfolitixorin works in a larger number of patients and has a stronger and longer efficacy in cancer treatment together with fluorouracil.

However, the efficacy of arfolitixorin has not yet been proven, and the substance has not been approved for the treatment of colorectal cancer. To date, arfolitixorin has been tested by around 420 volunteers and patients with colorectal cancer in different clinical studies. These studies have shown that arfolitixorin is safe and potentially can be of clinical benefit in patients with colorectal cancer when used in combination with fluorouracil, oxaliplatin and bevacizumab.

In the largest clinical study completed so far, arfolitixorin was shown to be equally effective compared to standard therapy with leucovorin, but not more effective. Additional results from this study suggested that the dose of arfolitixorin given did not deliver a sufficiently high amount of active substance into the tumor. Therefore, higher doses of arfolitixorin will be tested in this study to possibly achieve a better clinical effect. Further analyses also indicated that high accuracy regarding the timing and duration of the administration of the different treatments is important to achieve better efficacy of arfolitixorin.

Based on the available data, and the risk and benefit assessments performed, the Sponsor deems that it is relevant to further investigate the safety and tolerability, as well as the efficacy of arfolitixorin when given in combination with fluorouracil, oxaliplatin and bevacizumab. The proposed study design is believed to address all the main previous findings with the purpose to increase the efficacy with a remaining safety profile.

The study is divided into two parts. In the first part, up to five different doses of arfolitixorin will be investigated to find the optimal dose (i.e. the highest and well tolerated) of arfolitixorin as well as the optimal duration time of administration.

The second part of the study will be based on the results from the first part. Two doses of arfolitixorin will be tested for safety, tolerability and anti-tumor effect. In the second part, participants will be randomly assigned to one of two dose groups using a computer program. This so-called randomization procedure is comparable to tossing a coin.

All patients that participate in the study will receive treatment with arfolitixorin (+ fluorouracil, oxaliplatin and bevacizumab) every 2 weeks. The treatment will be given as an infusion into a vein. The number of treatment administrations that will be given is not predetermined but depends on the progression of the patient's disease.The treatment will continue every 2 weeks as long as the patient benefits from the treatment.

During the study period, the patient's disease and potential response to treatment, including shrinkage of the tumor and/or improvement of symptoms, will be monitored by imaging examinations, using so-called computer tomography (CT) or magnetic resonance imaging (MRI). The patient's state of health will also be monitored by physical examinations, and laboratory tests of urine and blood, as well as assessment of any side effects.

DETAILED DESCRIPTION:
This is a Phase 1b/2 study to determine the safety and preliminary efficacy of ARFOX + bevacizumab in patients with mCRC eligible for first-line therapy with 5-FU, oxaliplatin, and bevacizumab regimen. Prior treatment with 5-FU, oxaliplatin or bevacizumab administration for mCRC or more than 6 cycles (3 months) of oxaliplatin exposure during adjuvant treatment, is prohibited.

The study will include a Phase 1b dose-finding part followed by a randomized Phase 2 dose optimization part. Phase 1b will be conducted at 1 study site in Germany, and Phase 2 will be conducted at approximately 3 sites in Germany.

Eligible patients will undergo baseline assessments (within 28 days prior to treatment initiation) and repeat imaging using computed tomography (CT) or magnetic resonance imaging (MRI) after 6 and 12 weeks, and every 12 weeks thereafter as long as on study treatment.

All patients will receive treatment with ARFOX + bevacizumab every 14 days (+7 days) until progressive disease (PD), or clear clinical deterioration according to the Investigator's judgment, and as long as the patient is tolerating the treatment and agrees to continue.

After completion of study treatment, patients will complete an EOT visit within 30 days of discontinuation, and all patients should be followed in line with the site's standard of care scheme.

Subsequent study follow-up contacts/visits will be performed every 90 days (±15 days) after the EOT visit treatment, until 60% of the OS events have been collected or 24 months after last patient in (LPI), whichever comes first. The follow-up contacts may be conducted via telephone, via clinic visits, via local practitioner, via review of medical records or other means found suitable.

At the follow-up visits, information on any subsequent cancer treatments will be collected, recording and assessment of serious adverse events (SAEs) considered to be related to the study treatment will be performed, and survival status will be noted. All AEs collected during the reporting period still ongoing at the EOT visit will be followed until resolution or stabilization, or until deemed not necessary by the Investigator.

During the Phase 1b part of the study, a dose escalation design will be utilized to identify the optimal dose and duration of administration of arfolitixorin to be used in combination with 5-FU, oxaliplatin and bevacizumab. A Safety Review Committee (SRC) will review AEs, SAEs, dose-limiting toxicities (DLTs) and PK data and make recommendations regarding which dose level and cohort size to be tested for the next cohort, as well as the MTD. The SRC may also make recommendations of the duration of the infusion if there are safety findings that potentially correlate to a non-acceptable maximum plasma (peak) drug concentration (Cmax).

The dose escalation schema will be based on a Bayesian optimal interval (BOIN) design where the decision of dose escalation or de-escalation involves a simple comparison of the observed DLT rate at the current dose with the prespecified dose escalation and de-escalation boundaries.

The Phase 2 part of the study will be a randomized study where patients will be allocated to 1 of 2 dose levels of arfolitixorin, to be administered in combination with 5-FU, oxaliplatin and bevacizumab. The higher dose of arfolitixorin will be the MTD as determined in Phase 1b, and the lower dose will be a dose level below the MTD as determined in Phase 1b, i.e., 1 of the dose levels as determined by the SRC. The SRC will also review safety and efficacy data on a regular basis during Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF and ability to comply with protocol requirements.
* Histologically confirmed RAS mutant, MSS/pMMR, colorectal adenocarcinoma with metastatic disease, eligible for first-line therapy with 5-FU, oxaliplatin, and bevacizumab regimen.
* Tumor specimen (formalin-fixed, paraffin-embedded [FFPE]) available.
* Adequate heart function as defined as:

  1. Heart rate ≤100 bpm.
  2. Blood pressure ≤140/90.
  3. QTc ≤430 ms (males) or ≤450 ms (females).
  4. Ejection fraction (EF) >50%.
* Acceptable hematologic laboratory values defined as:

  1. Hemoglobin ≥90 g/L.
  2. Absolute neutrophil count ≥1.5 × 109/L.
  3. Platelets ≥100 × 109/L.
* Adequate organ function as defined by the following laboratory values:

  1. Total serum bilirubin ≤1.5 × upper limit of normal (ULN).
  2. ALT and AST ≤3 × ULN (≤5 × ULN in case of hepatic metastases).
  3. Creatinine ≤1.5 × ULN, or creatinine clearance ≥50 mL/min (as measured according to Cockcroft-Gault equation).
* Age ≥18 years at the time of signing the ICF.
* Radiographically measurable disease per RECIST (version 1.1) within 28 days of treatment allocation.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of >12 weeks.
* Female patients must be surgically sterile, postmenopausal, or have negative results for a pregnancy test at screening, on a serum or urine sample obtained within 72 hours prior to initiation of study treatment.
* Female patients of childbearing potential must agree to use highly effective contraceptive measures while on study treatment (ARFOX + bevacizumab) and for at least 15 months (or longer if according to local labels) after study treatment discontinuation. Highly effective methods are those that achieve a failure rate of less than 1% per year when used consistently and correctly (as per the Clinical Trial Coordination Group [CTCG] Recommendations related to contraception and pregnancy testing in clinical trials, Version 1.2, 07 Mar 2024).
* Female patients should agree to refrain from egg cell donation while on study treatment (ARFOX + bevacizumab) and for at least 15 months after the last dose of study treatment.
* Male patients with female partners of childbearing potential must agree to use adequate contraceptive measures while on study treatment (ARFOX + bevacizumab) and for at least 12 months (or longer if according to local labels) after study treatment discontinuation.
* Male patients should agree to refrain from sperm donation while on study treatment (ARFOX + bevacizumab) and for at least 12 months after the last dose of study treatment.

Exclusion Criteria:

* Indication for any mCRC surgery or anti-cancer treatment other than study treatment, including but not limited to resection as confirmed by a MTB.
* Concomitant malignancies or previous malignancies with less than a 2-year disease free interval at the time of signing consent. Patients with adequately treated basal or squamous cell carcinoma of the skin, or adequately treated carcinoma in situ (e.g., cervix) may enroll irrespective of the time of diagnosis. Patients with controlled, advanced prostate cancer are permitted. Ongoing adjuvant antihormonal therapy after breast or prostate cancer is permitted.
* Prior 5-FU, oxaliplatin or bevacizumab administration for mCRC. Or more than 6 cycles (3 months) of oxaliplatin exposure during adjuvant treatment.
* Known history of central nervous system (CNS) metastases or carcinomatous meningitis.
* Receipt of any investigational product within 14 days or 5 half-lives prior to study treatment initiation, whichever is shortest. Note that participation in any other clinical study is not allowed as long as the patient is on study treatment.
* Prior exposure to arfolitixorin.
* Major surgery, or significant traumatic injury within 8 weeks of study treatment initiation.
* Hypersensitivity to arfolitixorin, 5-FU, oxaliplatin or other platinum agent, or bevacizumab or to their excipients.
* Dihydropyrimidine dehydrogenase (DPD) enzyme deficiency test with a Clinical Pharmacogenetics Implementation Consortium (CPIC) activity score <1.
* Current evidence of any condition that makes participating in this study not in the best interest of the patient, including, but not limited to:

  1. Myocardial infarction or unstable angina within the past 6 months.
  2. New York Heart Association (NYHA) Class II or greater cardiac disease.
  3. Congestive heart failure.
  4. QT prolongation syndrome >430 ms (females) and >450 ms (males).
  5. Serious arrhythmias requiring medication for treatment.
  6. Active infection requiring i.v. antibiotics.
  7. Ongoing drug or alcohol abuse.
* Sensory peripheral neuropathy Grade ≥2.
* Pregnancy or lactation.
* Any medical condition, which in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities, or any psychological, familial, sociological or geographical condition that potentially hampers compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: To evaluate the safety and tolerability of ARFOX + bevacizumab in patients with mCRC. | From enrollment until end of study, i.e. until death, an average of 24 months.
  To evaluate the safety and tolerability of ARFOX + bevacizumab in patients with mCRC, by measuring number and severity of AEs and clinically significant abnormal laboratory findings, regardless of causal relationship to ARFOX + bevacizumab. The outcome of Phase 1b is to determine the MTD of arfolitixorin (ARFOX + bevacizumab) in patients with mCRC.
Phase 2: To evaluate the safety and tolerability of two pre-defined doses of arfolitixorin (MTD and a dose level below MTD; ARFOX + bevacizumab) in patients with mCRC. | From enrollment until end of study, i.e. until death, an average of 24 months.
  To evaluate the safety and tolerability of two pre-defined doses of arfolitixorin (MTD and a dose level below MTD; ARFOX + bevacizumab) in patients with mCRC, by measuring number and severity of AEs, including clinically significant abnormal laboratory findings, regardless of causal relationship to ARFOX + bevacizumab.
Phase 2: To assess the anti-tumor activity of arfolitixorin (MTD and a dose level below MTD; ARFOX + bevacizumab) in patients with mCRC, in terms of ORR. | From enrollment until end of treatment, i.e. until progressive disease, or clear clinical deterioration according to the Investigator's judgment, and as long as the patient is tolerating the treatment and agrees to continue, an average of 11 months.
  To assess the anti-tumor activity of arfolitixorin (MTD and a dose level below MTD; ARFOX + bevacizumab) in patients with mCRC, in terms of ORR, defined as the proportion of patients who have BOR of CR, or PR, measured by RECIST (version 1.1).

SECONDARY OUTCOMES:
Phase 1b: To assess the anti-tumor activity of ARFOX + bevacizumab in patients with mCRC in terms of ORR | From enrollment until end of treatment, i.e. until progressive disease, or clear clinical deterioration according to the Investigator's judgment, and as long as the patient is tolerating the treatment and agrees to continue, an average of 11 months.
  To assess the anti-tumor activity of ARFOX + bevacizumab in patients with mCRC in terms of ORR, defined as the proportion of patients who have BOR of CR, or PR, measured by RECIST (version 1.1).
Phase 1b: To assess the anti-tumor activity of ARFOX + bevacizumab in patients with mCRC in terms of PFS. | From the first study dose date to the date of first documentation of disease progression or death (whichever occurs first), an average 11 months.
  To assess the anti-tumor activity of ARFOX + bevacizumab in patients with mCRC in terms of PFS, defined as the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurs first).
Phase 1b: To assess the anti-tumor activity of ARFOX + bevacizumab in patients with mCRC in terms of OS. | From enrollment until end of study, i.e. until death, an average of 24 months.
Phase 1b: To determine the PK profile of arfolitixorin, administered in combination with oxaliplatin and 5-FU. | Assessed just before the end of the infusion of arfolitixorin, and at 5, 10, 20, and 60 minutes after finished infusion of arfolitixorin, on day 1 and day 15..
  To determine the PK profile of arfolitixorin, administered in combination with oxaliplatin and 5-FU, by measuring plasma concentration of arfolitixorin
Phase 2: To assess the anti-tumor activity of arfolitixorin (MTD and a dose level below MTD; ARFOX + bevacizumab) in patients with mCRC, in terms of OS. | From enrollment until end of study, i.e. until death, an average of 24 months.
Phase 2: To assess the anti-tumor activity of arfolitixorin (MTD and a dose level below MTD; ARFOX + bevacizumab) in patients with mCRC, in terms of PFS. | From the first study dose date to the date of first documentation of disease progression or death (whichever occurs first), an average 11 months.
  To assess the anti-tumor activity of ARFOX + bevacizumab in patients with mCRC in terms of PFS, defined as the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Stintzing, Prof. Dr. MD, Principal Investigator — Charité - Universitaetsmedizin Berlin, Berlin, 10117
Locations (1):
- Charité - Universitaetsmedizin Berlin, Berlin, Germany